CLINICAL TRIAL: NCT06484049
Title: Prospective Observational Clinical Study on Changes in Cognitive Levels in Elderly Patients Before and After Hematopoietic Stem Cell Transplantation
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: IIT2024042
Record Dates: First submitted 2024-06-06; First posted 2024-07-03 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-06

CONDITIONS: Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the potential improvement in cognitive levels in elderly individuals following hematopoietic stem cell transplantation, which will help better understand the changes in cognitive levels after transplantation in elderly patients, providing crucial reference for future clinical practice and research.

DETAILED DESCRIPTION:
To investigate the potential improvement in cognitive levels in elderly individuals following hematopoietic stem cell transplantation, which will help better understand the changes in cognitive levels after transplantation in elderly patients, providing crucial reference for future clinical practice and research.

To observe changes in cognitive levels in patients aged ≥55 years receiving allogeneic hematopoietic stem cell transplantation (allo-HSCT) before and after allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 55 years;
2. Patients planning to undergo allogeneic hematopoietic stem cell transplantation.

Exclusion Criteria:

1. Patients with active diseases;
2. Presence of central nervous system tumor invasion;
3. Planning to undergo two or more transplantations;
4. Severe cognitive impairments or mental illnesses;
5. Inability to communicate in Mandarin.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age greater than or equal to 55 years; Patients planning to undergo allogeneic hematopoietic stem cell transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
To observe changes in cognitive levels in patients aged ≥55 years receiving allogeneic hematopoietic stem cell transplantation (allo-HSCT) before and after allo-HSCT. | 1YEAR
  1.Post-transplant Assessment: Cognitive level follow-up assessments at 1 month, 3 months, 6 months, and 1 year post-operation. Evaluation content is consistent with pre-transplant assessments. Cerebrospinal fluid testing is scheduled for 3 months post-transplant.4. Survival and Disease Follow-up: Follow-up for one year after transplantation to observe overall survival rate, disease-free survival rate, etc.

IPD SHARING:
Plan to Share IPD: No